CLINICAL TRIAL: NCT07298148
Title: A Multicenter, Prospective, Phase II, Single-Arm Study of Firmonertinib 160 mg in Patients With EGFR-Mutant Advanced NSCLC Demonstrating Stable Disease After 8 Week Induction With Firmonertinib 80 mg
Brief Title: Firmonertinib 160 mg in Patients With EGFR-Mutant Advanced NSCLC Demonstrating SD After 8 Week Induction With Firmonertinib 80 mg
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025YJZ88
Record Dates: First submitted 2025-12-11; First posted 2025-12-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: NSCLC Stage IV; EGFR Positive Non-small Cell Lung Cancer; EGFR-TKI Sensitizing Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Firmonertinib 160mg (Experimental)
  Interventions: Drug: Firmonertinib 160mg

INTERVENTIONS:
Drug: Firmonertinib 160mg — Patients enter an 8-week induction phase at 80 mg once daily. Those with stable disease per RECIST v1.1 at Week 8 escalate to 160 mg daily until disease progression or unacceptable toxicity.

SUMMARY:
This study evaluates the efficacy and safety of Firmonertinib 160 mg once daily in patients with EGFR-mutant, advanced NSCLC who achieve stable disease after first-line Firmonertinib 80 mg for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years.
* ECOG performance status 0-1; life expectancy ≥3 months.
* Histologically/cytologically confirmed advanced/metastatic non-squamous NSCLC unsuitable for curative therapy.
* Documented EGFR 19del or L858R mutation.
* No prior systemic therapy for advanced disease.
* Stable disease after 8 weeks of Firmonertinib 80 mg daily.
* more than 1 measurable lesion per RECIST v1.1.
* Adequate hematologic, renal, hepatic, and coagulation function.
* Signed written informed consent.

Exclusion Criteria:

* Hypersensitivity to Firmonertinib or related compounds.
* Other actionable oncogenic drivers (ALK, ROS1, RET, BRAF, NTRK, MET, KRAS, except TP53/RB1).
* Prior EGFR-TKI therapy or prohibited concomitant medications.
* Unresolved toxicities >CTCAE Grade 1 (except allowed conditions).
* Symptomatic CNS metastases or spinal cord compression.
* GI disorders impairing drug absorption.
* Uncontrolled systemic diseases or active infections (HBV/HCV/HIV).
* Interstitial lung disease (history or active).
* Clinically significant cardiac abnormalities including QTc >470 ms or LVEF <50%.
* Pregnancy or breastfeeding.
* Any condition compromising compliance.
* CR, PR, or PD at completion of induction therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From dose escalation (Week 8) until documented disease progression or start of new anticancer therapy, assessed approximately every 8 weeks, up to 24 months.
  Percentage of patients achieving CR or PR per RECIST v1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From first dose to disease progression or death, whichever occurs first; followed for up to 24 months.
  Time from the start of randomization (or the start of treatment in a single-arm trial) to tumor progression or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | From dose escalation (Week 8) until documented disease progression or start of new anticancer therapy, assessed approximately every 8 weeks, up to 24 months.
  Percentage of patients achieving CR, PR, or SD.per RECIST v1.1.
Duration of Response (DoR) | From dose escalation (Week 8) until documented disease progression or start of new anticancer therapy, assessed approximately every 8 weeks, up to 24 months.
  Duration from first response to progression or death.
CNS Objective Response Rate (CNS-ORR) | From dose escalation (Week 8) until documented disease progression or start of new anticancer therapy, assessed approximately every 8 weeks, up to 24 months.
  Evaluated via CNS imaging per RECIST v1.1 or applicable CNS criteria.
Incidence of Treatment-related adverse event (TRAE) | From first dose of therapy through 30 days after last dose of study treatment up to 24 months.
  any adverse event that in the investigator's opinion may have been caused by the study medication with reasonable possibility per CTCAE 5.0.

IPD SHARING:
Plan to Share IPD: No